CLINICAL TRIAL: NCT05673278
Title: To Examine the Feasibility of Non-Invasive Monitoring With Bowel Ultrasound in Paediatric Inflammatory Bowel Disease and Correlation With Inflammatory Markers, Disease Activity Scores and as a Predictor of Changes in Treatment (NIMBUS)
Brief Title: Non-Invasive Monitoring Through Bowel Ultrasound in Paediatric Inflammatory Bowel Disease Study
Acronym: NIMBUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Other Study IDs: 8497/OCT/2022
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2022-11

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease; Pediatric Crohns Disease; Pediatric Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease; Pediatric ulcerative colitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and young people diagnosed with inflammatory bowel disease aged 2-19 years: Diagnosis according to the modified Porto criteria All participants will undergo single ultrasound scan which will be evaluated with medical notes and results from routine care. No new samples will be taken outside of normal care.
  Interventions: Diagnostic Test: Bowel Ultrasound Scan

INTERVENTIONS:
Diagnostic Test: Bowel Ultrasound Scan — Ultrasound scans will attempt to measure predefined criteria implemented in other research work using bowel ultrasound.
  I - Bowel wall thickness II - Colour Doppler signal III - Loss of wall layer stratification IV - Loss of haustration V - Fatty wrapping VI - Motility in terminal ileum (TI) VII - Lymphadenopathy VIII - Abscess IX - Stricture
  + Image quality

SUMMARY:
Rates of inflammatory bowel disease (IBD) are increasing rapidly in children and young people, and targets for management are becoming more demanding, with better control of disease to prevent complications, cancers and surgeries. This project "Non-Invasive Monitoring Through Bowel Ultrasound in Paediatric Inflammatory Bowel Disease" or NIMBUS study will aim to explore the possibility of using ultrasound to examine inflammation in this group.

Monitoring inflammation in this population currently is done with regular endoscopy (camera tests) and/ or MRI enterography scans which are invasive, can be uncomfortable, expensive and may have long waiting lists. These studies also require bowel prep, in the form of laxative medicines which can be distressing and cause time off from school. Direct visualisation through ultrasound could allow better monitoring of disease, and is quick, accurate, non-invasive and relatively low-cost. This could also allow for more appropriate medication use and a decrease in over/under use of medicines.

This study will aim to recruit 50 children and young people with inflammatory bowel disease. Each child will have an ultrasound scan after enrolment and the investigators will use the information from these scans, as well as routine blood tests (already taken in normal care) and follow up medical information to explore the use of ultrasound in this group. The investigating team will aim to contribute to the global discussion around this topic and if results are positive will aim to improve monitoring for this population managed at the Noah's Ark Children's Hospital for Wales.

DETAILED DESCRIPTION:
This research project will aim to examine the use of ultrasound scans for monitoring disease in paediatric patients with inflammatory bowel disease. This is an area which is being explored in adult research, however it is under-utilised in children and young people.

The null hypothesis in this study is that there is no association between gut ultrasound findings and blood and stool tests of inflammation or disease activity scores in paediatric patients with inflammatory bowel disease. The alternative hypothesis is that there is an association between ultrasound findings and these parameters. Regarding the follow up part of the study, the null hypothesis is that abnormal ultrasound findings have no correlation with either increase or decrease in treatment. The alternative hypothesis is that abnormal ultrasound findings correlate with increase in treatment and normal findings with no change or decrease in treatment.

A prospective feasibility observational methodology will be employed.

In terms of timetable for the study, preparation, including seeking of ethical and research and development alongside study logistics will be undertaken in the first 3 months. Participants will be recruited between months 4 and 18, with data collection and assessment over this time frame. Data will be analysed from months 6 to 24.

Recruitment of children will occur at a routine point of contact with paediatric gastroenterology services, i.e. inpatient review, outpatient attendance for infusion, clinic appointment or endoscopy, or through a virtual recruitment process, where deemed appropriate by the study team. Participants and their families will be provided with age-appropriate information and offered time to review these resources before obtaining consent. When recruited, study team will collect initial recruitment data, i.e. baseline characteristics. The investigating team will aim to arrange for ultrasound appointment as part of routine visit or during inpatient admission. On the day of ultrasound participants will attend the Noah's Ark children's hospital for Wales and scan will be undertaken. The trial team will review recent results (routine tests taken as part of normal care) at this point and then medical notes for clinical outcome up to twelve months after the scan. Results of project will be fed back to participants after study closure.

This project will be open to children with a diagnosis of IBD, according to the modified Porto criteria, aged between 2-19 years old. Only children without these diagnoses, those who have had surgery, which could act as a potential confounder in ultrasound findings, those outside of the age range and those belonging to families unable to give informed consent will be excluded. The information recorded from ultrasound scans will not be made available to the clinical team, therefore recruitment biases will be minimised. The target sample size of 50 children and young people has been set to achieve meaningful results and minimise statistical error. This figure is also based on other fledgling work in this area.

ELIGIBILITY:
Inclusion Criteria:

* 50 children visiting hospital for clinical appointments (clinic, infusions, endoscopy etc.) or inpatient in hospital with flare of disease.
* Children with IBD, aged 2-19 years, diagnosed according to the modified Porto criteria

Exclusion Criteria:

* Children who do not have inflammatory bowel disease
* Patients who have previously undergone bowel resection (subtotal colectomy, right hemicolectomy or stricturoplasty)
* Patients or families unable to give informed consent
* Children under 2 years of age or patients older than 19 years

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young people with inflammatory bowel disease under the care of Noah's Ark Children's Hospital for Wales
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility metrics (recruitment, retention/follow up) | 12-24 months
  Reported as point estimates alongside 95% CIs, and assessed against the traffic light progression criteria:
  * Recruitment rate (number screened and approached / number consented): >60% green, 30-60% amber, <30% red
  * Retention/follow up rate (number consented / number providing outcome data): >80% green, 70-80% amber, <70% red
  * Availability rate of ultrasound scan attendance and specific parameters i.e. ability to obtain for example "loss of bowel wall haustrations" (number scanned/ number providing outcome data): >80% green, 70-80% amber, <70% red
Ultrasound parameter score total | 12-24 months
  Composite measure of bowel wall thickness (BWT), colour doppler signal, loss of wall layer stratification, loss of haustration, fatty wrapping, motility in TI, lymphadenopathy and abscess/ stricture. Bowel wall thickness will be defined as thickness in longitudinal plane + thickness in cross-sectional plane with the total being divided by 2. BWT > 3.0 mm for colonic segments and BWT > 2.0 mm for terminal ileum will be considered abnormal. Colour doppler signal will be graded from 0 to 3. All other parameters are binary and will be scored as either 0 (absent) or 1 (present). A total score will make up the primary outcome measure. Correlations with routine measures of inflammation (i.e blood tests and disease activity scores will be explored).

SECONDARY OUTCOMES:
Increase or decrease in medical management | 12 months
  Recorded from medical notes up to 12 months post ultrasound scan. Defined as increase, decrease or remaining unchanged.
Complications | 12 months
  Recorded from medical notes up to 12 months post ultrasound scan. Recording of surgeries, admissions or flare of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Martin O Edwards, PhD FRCPCH, Principal Investigator — Cardiff and Vale University Health Board
Locations (1):
- Noah's Ark Children's Hospital for Wales, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Green Z, Towriss C, Ashton JJ, Beattie RM, Evans A, Wahid A, Edwards M. Noninvasive monitoring with bowel ultrasound (NIMBUS) in paediatric inflammatory bowel disease: Feasibility in a single centre. J Pediatr Gastroenterol Nutr. 2025 Oct;81(4):1014-1023. doi: 10.1002/jpn3.70159. Epub 2025 Jul 21. PMID 40686225
- [Derived] Green Z, Mayberry E, Ashton JJ, Beattie RM, Evans A, Wahid A, Edwards MO. NIMBUS study protocol: a single-centre feasibility study of non-invasive monitoring with bowel ultrasound in paediatric inflammatory bowel disease. BMJ Open. 2023 Dec 14;13(12):e078675. doi: 10.1136/bmjopen-2023-078675. PMID 38101846